CLINICAL TRIAL: NCT06856616
Title: Machine Learning Models for Predicting Long-Term Clinical Outcomes in Chinese Female Breast Cancer Patients Receiving Neoadjuvant Chemotherapy
Brief Title: Predicting Long-Term Clinical Outcomes in Chinese Breast Cancer Patients Receiving Neoadjuvant Chemotherapy
Status: Active, not recruiting | Type: Observational
Sponsor: The Third Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Ming Niu, Prof., The Third Affiliated Hospital of Harbin Medical University
Other Study IDs: MNiu
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-02

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Harbin Medical University Cancer Hospital
- Quanzhou First Hospital Affiliated to Fujian Medical University
- Xiamen Maternity and Child Healthcare Hospital

SUMMARY:
At present, the majority of studies on neoadjuvant chemotherapy (NAC) in patients with breast cancer (BC) use pathological complete response (pCR) as a surrogate marker for patient prognosis, with significant improvements in pCR indicating better long-term survival. However, there is still a lack of non-invasive tools for accurately predicting the prognosis and pCR of BC patients undergoing NAC. Recent research has introduced emerging artificial intelligence machine learning (ML) and deep learning (DL) algorithms such as Bayesian methods, K-nearest neighbors (KNN), decision trees, support vector machines (SVM), XGBoost, ResNet, convolutional neural networks, and Transformer models, which have brought new avenues of exploration for cancer researchers.

The integration of AI with imaging, pathology, genomics, and other multi-omics has non-invasively improved preoperative diagnosis of breast cancer and, when combined with clinical factors, can assess postoperative survival. Moreover, current research data is limited, and reliable predictive models require extensive data for training. Therefore, establishing a multi-center database is essential.

ELIGIBILITY:
Inclusion Criteria:

1. Women with invasive breast cancer who received neoadjuvant chemotherapy (NAC) treatment in various hospitals from 2008 to 2019 (follow-up endpoint December 31, 2024)
2. Women with primary breast cancer (Stage II-III) confirmed by pre-NAC needle biopsy, along with recorded clinical, pathological, and prognostic information
3. With MR images before the first cycle of NAC and before surgery
4. With pathological HE staining images, including biopsy pathology and postoperative major pathology

Exclusion Criteria:

1. Any form of treatment was received before NAC, including endocrine therapy, radiotherapy, and chemotherapy
2. Disease metastasis occurred during NAC
3. Breast cancer patients with secondary malignancies from other cancers
4. Patients did not complete surgery and were lost to follow-up

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From 2008 to 2019 (with follow-up ending on December 31, 2024), women with invasive breast cancer who received NAC treatment at various hospitals
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
5-10 year survival rate | 2008-2019
  5-10 year survival rate of female breast cancer patients treated with neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Ming Niu, Harbin, Longjiang Hei, China

IPD SHARING:
Plan to Share IPD: No
Reasonable needs can be in contact with the research head